CLINICAL TRIAL: NCT00034541
Title: Phase Ib/IIa Study of an Anti-Epidermal Growth Factor Receptor (EGFr) Antibody Cetuximab in Combination With Carboplatin-Paclitaxel in Patients With Chemotherapy-Naive Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Cetuximab in Combination With Carboplatin-Paclitaxel in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: University of Colorado, Denver (Other); Greenwich Hospital (Other); Indiana University (Other)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP02-9932
Record Dates: First submitted 2002-04-30; First posted 2002-05-01 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: cetuximab; epidermal growth factor receptor; antibody; non-small cell lung cancer; carboplatin; paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): An initial dose of cetuximab (400 mg/m2 i.v. over 120 minutes) will be administered 1 week prior to the initiation of chemotherapy. Thereafter, cetuximab will be infused weekly at maintenance doses of 250 mg/m2 (over 60 minutes). On the first day of each cycle (every 3 weeks) of therapy, a 3-hour paclitaxel (225 mg/m2) infusion will be administered 1-hour post completion of the cetuximab infusion, immediately followed by a 30-minute carboplatin (AUC=6) infusion.
  Interventions: Biological: cetuximab; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Biological: cetuximab — 400 mg/m2 i.v. over 120 minutes
  Other Names: Erbitux
Drug: paclitaxel — 225 mg/m2, infusion
  Other Names: Taxol
Drug: carboplatin — 30-minute AUC = 6, infusion.
  Other Names: Paraplatin

SUMMARY:
The study will enroll approximately 33 EGFr positive chemotherapy-naive stage IV non-small cell lung cancer patients. Patients will receive cetuximab in combination with carboplatin and paclitaxel for two cycles or until disease progression or until the patient exhibits intolerable toxicities. Patients will be evaluated for efficacy and safety throughout the duration of the study.

DETAILED DESCRIPTION:
The study will enroll approximately 33 chemotherapy-naive stage IV non-small cell lung cancer patients. Patients will receive 3-week cycles of therapy with the exception of the initial cycle where the patients will receive 4 cycles of therapy. Patients will be enrolled after EGFr expression is confirmed and the study inclusion and exclusion criteria are met. An initial dose of cetuximab will be administered prior to the initiation of chemotherapy. Thereafter, cetuximab will be infused weekly. On the first day of each cycle, a paclitaxel infusion will be administered post completion of the cetuximab infusion, immediately followed by a carboplatin infusion. Patients will receive cetuximab in combination with carboplatin and paclitaxel for two cycles or until disease progression or until the patient exhibits intolerable toxicities. Patients will be evaluated for a tumor response at the end of every two cycles of therapy and evaluated for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria must be met:

* The patient has stage IV NSCLC with either present or prior histologic or pathologic confirmation of NSCLC
* The patient has uni-dimensionally measurable stage IV NSCLC
* The patient has chemotherapy-naive stage IV NSCLC. The patient may have recurrent disease if prior radiation therapy was received. Pathological confirmation of recurrence is required for disease within a radiation portal.
* The patient's ECOG performance status is ≤ 2 at study entry.
* The patient has immunohistochemical evidence of EGFr expression (≥1+). Patients who do not have tumor tissue available for EGFr testing will undergo a biopsy of an accessible tumor. EGFr expression must be confirmed prior to study entry.
* The patient has given signed informed consent.
* The patient is 18 years of age or older.
* The patient has adequate hematologic function, as defined by an absolute neutrophil (ANC)≥ 1,500/mL3 , a WBC count≥3,000/mL3, a platelet count ≥100,000/mL3, and a hemoglobin level ≥9g/dL.
* The patient has adequate hepatic function as defined by a total bilirubin level ≤1.5 X the upper limit of normal (ULN) and an alkaline phosphatase, AST, and ALT level ≤2.5 X the ULN.
* The patient has adequate renal function with a serum creatinine level ≤1.5 mg/dL or a creatinine clearance ≥60 cc/minute.
* The patient is disease free from a previously treated malignancy, other than the disease under study, for greater than 3 years (patients with a history of a previous basal cell carcinoma of the skin or preinvasive carcinoma of the cervix will not be excluded).
* The patient, if a woman, agrees to use effective contraception if childbearing potential exists. The patient, if a man, agrees to use effective contraception.

Exclusion Criteria:

The following ten exclusion criteria are for this study:

* The patient has received prior cetuximab therapy.
* The patient has disease amenable to curative surgery.
* The patient has received prior chemotherapy for the disease under study.
* The patient has received wide field radiation therapy within 4 weeks prior to the first infusion of cetuximab. The patient may have local irradiation for the management of tumor-related symptoms.
* The patient has undergone major thoracic or abdominal surgery within 30 days (to allow for a full recovery)prior to the first infusion of cetuximab.
* The patient has a history of uncontrolled angina,arrhythmias, or congestive heart failure.
* The patient has uncontrolled seizure disorder, active neurological disease (not tumor related), or grade ≥2 neuropathy (patients with meningeal or central nervous system [CNS] involvement by the tumor will be eligible).
* The patient has a history of hypersensitivity to Cremophor EL.
* The patient, if a woman, is pregnant (confirmed by serum BHCG) or breastfeeding.
* The patient has received any investigation agents within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-12; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of cetuximab when used in combination with paclitaxel and carboplatin | 8 Weeks

SECONDARY OUTCOMES:
Antitumor activity | 8 Weeks
Effect of cetuximab on the pharmacokinetics of paclitaxel and carboplatin | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (3):
- United States (3):
  - ImClone Investigational Site, Denver, Colorado
  - ImClone Investigational Site, Greenwich, Connecticut
  - ImClone Investigational Site, Indianapolis, Indiana

REFERENCES:
- [Result] Thienelt CD, Bunn PA Jr, Hanna N, Rosenberg A, Needle MN, Long ME, Gustafson DL, Kelly K. Multicenter phase I/II study of cetuximab with paclitaxel and carboplatin in untreated patients with stage IV non-small-cell lung cancer. J Clin Oncol. 2005 Dec 1;23(34):8786-93. doi: 10.1200/JCO.2005.03.1997. Epub 2005 Oct 24. PMID 16246975
- [Result] Kelly K, Hanna N, Rosenberg A, Bunn PA, Needle MN. A multi-centered phase I/II study of cetuximab in combination with paclitaxel and carboplatin in untreated patients with stage IV non-small cell lung cancer (Abstract 2592). American Society of Clinical Oncology Annual Meeting. 2003 May 31-June 3; Chicago, Illinois.